## **Statistical Analysis Plan**

Study Title: Long-term Telerehabilitation for Patients With Stroke

ClinicalTrials.gov Identifier: NCT03460587

November 22, 2020

**Statistical analysis plan**: Data analysis used non-parametric statistical testing (JMP 13, SAS; Cary, NC). All analyses were two-tailed, with statistical significance set at p<0.05 and no corrections made for multiple comparisons in this feasibility study.